CLINICAL TRIAL: NCT01004731
Title: Phase Ib, IIa Study of Anti-Epidermal Growth Factor Receptor (EGFr) Antibody, Cetuximab, in Combination With Gemcitabine/Carboplatin in Patients With Chemotherapy-Naive Stage IV Non-Small Cell Lung Cancer
Brief Title: Study of Anti-Epidermal Growth Factor Receptor (EGFr) Antibody, Cetuximab, in Combination With Gemcitabine/Carboplatin in Patients With Stage IV Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Michael James Bertram, Proffessor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X010524006; UAB 9909 (Other: UAB Department study number); NCT00027755 (obsolete NCT alias)
Record Dates: First submitted 2009-10-21; First posted 2009-10-30 (Estimated); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Stage IV Non-Small Cell Lung Cancer
Keywords: EGFr; cetuximab; gemcitabine; carboplatin; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab in combination with Carboplatin/Gemcitabine (Experimental): Approximately 30 patients with advanced NSCLC will be enrolled. Patients will receive 3-week cycles of Cetuximab in combination with Carboplatin/Gemcitabine.
  Interventions: Drug: Cetuximab in combination with Carboplatin/Gemcitabine

INTERVENTIONS:
Drug: Cetuximab in combination with Carboplatin/Gemcitabine — A loading dose of Cetuximab (400 mg/m2 IV over 120 minutes) will be administered 1 week prior to chemotherapy. Thereafter, Cetuximab will be infused weekly at maintenance doses of 250 mg/m2 (over 60 minutes). On the first day of each new cycle of therapy, Carboplatin will be infused with Gemcitabine (Days 1 and 8). Patients will be evaluated for a tumor response following every two cycles of therapy. In the absence of progressive disease, patients may continue to receive additional therapy.

SUMMARY:
The objective is to evaluate the toxicity profile, response rate, and time to progression of Cetuximab administered in combination with either Carboplatin + Gemcitabine in patients with advanced non-small cell lung cancer with positive EGFr expression.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety profile of Cetuximab when used in combination with gemcitabine and carboplatin in patients with EGFr positive, chemotherapy-naive, stage IV non-small cell lung cancer (NSCLC).

Also, the study will determine the response rate in patients with EGFr positive chemotherapy-naive, stage IV non-small cell lung cancer (NSCLC) treated with Cetuximab in combination with gemcitabine and carboplatin as well as determine the time to progression in patients with EGFr positive chemotherapy-naive, stage IV NSCLC treated with Cetuximab in combination with gemcitabine and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of histologically/cytologically confirmed advanced non- small cell lung cancer (NSCLC).
* Have uni-dimensionally measurable and/or evaluable advanced NSCLC.
* Have Stage IV or recurrent disease following radiation therapy.
* Have ECOG performance status of 0-1 or Karnofsky performance status of 80- 100 at study entry.
* Have given signed informed consent.
* Be at least 18 years of age.
* Have ANC greater than or equal to 1,500/mm3, platelets greater than or equal to 100,000/mm3, WBC greater than or equal to 3,000 mm3, and hemoglobin greater than or equal to 9 g/dL.
* Have total bilirubin less than or equal to 1.5 x upper limits of normal, Alk Phos, AST and ALT less than or equal to 2.5 x upper limits of normal.
* Have serum creatinine less than or equal to 1.5 mg/dL, or calculated creatinine clearance greater than or equal to 60 cc/minute.
* Be disease free from a previously treated malignancy for more than three years. Patients with a history or a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix will not be excluded.
* Agree to use effective contraception if procreative potential exists.
* Must have positive EGFr expression (tumor tissue) by immunohistochemical assay.

Exclusion Criteria:

* Have received prior murine monoclonal antibody or Cetuximab therapy.
* Have disease amenable to curative surgery.
* Have received prior chemotherapy.
* Have received radiation therapy within 3 weeks prior to the first infusion of Cetuximab.
* Have a history of clinically significant cardiac disease, serious arrhythmias, or significant conduction abnormalities, in the judgment of the PI.
* Have uncontrolled seizure disorder, active neurological disease, or Grade 2 or higher neuropathy.
* Be pregnant or breast-feeding.
* Have received any investigational agent(s) within 1 month of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-06; Primary Completion 2002-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the tumor response of cetuximab in combination with gemcitabine and carboplatin in patients with EGFr positive, chemotherapy-naive, Stage IV non-small cell lung cancer. | 3-week cycles with evaluation after every 2 cycles until disease progression or unacceptable toxicity

SECONDARY OUTCOMES:
Evaluate the response rate and time to disease progression | 3-week cycles with evaluation after every 2 cycles until disease progression or unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States